CLINICAL TRIAL: NCT02859467
Title: Benefits of Kinesio Taping and Inhibitory Treatment Techniques in Patients With Fibromyalgia Syndrome
Brief Title: Kinesio Taping and Inhibitory Treatment Techniques
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Adelaida María Castro-Sánchez, Professor, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UAL-496
Record Dates: First submitted 2016-08-04; First posted 2016-08-09 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Fibromyalgia
Keywords: Physical Therapy Modalities; Exercise; Electrical Stimulation Therapy; Bandages
MeSH Terms: conditions — Fibromyalgia; Motor Activity | interventions — Exercise; Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kinesio Taping and Inhibitory Treatment Techniques (Experimental): During each session participants will receive the application kinesio taping in trapezius, infraspinatus and paravertebral muscles.
  Inhibitory Treatment Techniques:
  * Release Technique of the trapezius muscle.
  * Release Technique for scalene muscles.
  * Technique suboccipital inhibition.
  * Technique hands crossed for induction dorsal superficial fascia.
  Interventions: Other: Kinesio Taping and Inhibitory Treatment Techniques
- Exercise and Electrical Stimulation Therapy (Active Comparator): Session for general physical activities (joint mobility, muscle strength and elasticity), and electrical stimulation therapy on para vertebral muscles.
  Interventions: Other: Exercise and Electrical Stimulation Therapy

INTERVENTIONS:
Other: Kinesio Taping and Inhibitory Treatment Techniques — Kinesio Taping on trapezius, infraspinatus, and paravertebral muscles
  Inhibitory Treatment Techniques:
  * Release Technique of the trapezius muscle.
  * Release Technique for scalene muscles.
  * Technique suboccipital inhibition.
  * Technique hands crossed for induction dorsal superficial fascia.
  Arms: Kinesio Taping and Inhibitory Treatment Techniques
Other: Exercise and Electrical Stimulation Therapy — Session for general physical activities (joint mobility, muscle strength and elasticity), and electrical stimulation therapy on para vertebral muscles.
  Arms: Exercise and Electrical Stimulation Therapy

SUMMARY:
Objective: Compare the benefits of Kinesio Taping and Inhibitory Treatment Techniques for Cervical, Thoracic and Lumbar Spine in Patients with Fibromyalgia Syndrome (FMS).

Study Design: A single-blind randomized controlled trial was conducted on patients with FMS.

Setting: Clinical setting. Methods: Sixty-four subjects with FMS were randomly assigned to an experimental group receiving kinesio taping and inhibitory treatment techniques, or to a control group for exercises and electrical stimulation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Fibromyalgia Syndrome.
* Limitation of usual activities due to pain on at least 1 day in the previous 30 days.
* Agreement to attend evening therapy sessions.
* Non-practice of regular physical activity.

Exclusion Criteria:

* A history of surgery.
* The presence of comorbid conditions (e.g., morbid obesity, inflammatory diseases, irritable bowel syndrome and interstitial cystitis).
* A history of whiplash injury.
* Severe physical disability.
* uncontrolled endocrine disorders (e.g., hyperthyroidism, diabetes); 6) illness (e.g., schizophrenia or substance abuse).
* The use of medication other than as-needed analgesics (excluding long-term narcotics).
* Malignancy.
* Psychiatric disorders.
* A score of ≥ 9 points in the Beck depression inventory.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Changes from Baseline, and 10 weeks
  A 10-point Numerical Pain Scale (0: no pain, 10: maximum pain) assesses the intensity of pain.

SECONDARY OUTCOMES:
Quality of Life (SF-36) | Changes from Baseline, and 10 weeks
Pittsburgh Quality of Sleep Questionnaire | Changes from Baseline, and 10 weeks
Beck Inventory for Depression | Changes from Baseline, and 10 weeks
Fibromyalgia Impact Questionnaire (FIQ) | Changes from Baseline, and 10 weeks
Hospital Anxiety Depression Scale (HADS) | Changes from Baseline, and 10 weeks
State-Trait Anxiety Inventory (STAI) | Changes from Baseline, and 10 weeks
McGill Pain Questionnaire | Changes from Baseline, and 10 weeks
Fatigue Impact Scale | Changes from Baseline, and 10 weeks
Pain Pressure | Changes from Baseline, and 10 weeks
Schöber Test | Changes from Baseline, and 10 weeks
Widespread pain index | Changes from Baseline, and 10 weeks
Symptom severity score | Changes from Baseline, and 10 weeks
Measurement Finger-Floor | symptom severity scale

CONTACTS AND LOCATIONS:
Locations (1):
- Adelaida María Castro-Sánchez, Almería, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Macfarlane GJ, Kronisch C, Dean LE, Atzeni F, Hauser W, Fluss E, Choy E, Kosek E, Amris K, Branco J, Dincer F, Leino-Arjas P, Longley K, McCarthy GM, Makri S, Perrot S, Sarzi-Puttini P, Taylor A, Jones GT. EULAR revised recommendations for the management of fibromyalgia. Ann Rheum Dis. 2017 Feb;76(2):318-328. doi: 10.1136/annrheumdis-2016-209724. Epub 2016 Jul 4. PMID 27377815
- [Background] Fernandez-de-Las-Penas C, Arendt-Nielsen L. Myofascial pain and fibromyalgia: two different but overlapping disorders. Pain Manag. 2016 May;6(4):401-8. doi: 10.2217/pmt-2016-0013. Epub 2016 Jun 14. PMID 27296946
- [Background] Saral I, Sindel D, Esmaeilzadeh S, Sertel-Berk HO, Oral A. The effects of long- and short-term interdisciplinary treatment approaches in women with fibromyalgia: a randomized controlled trial. Rheumatol Int. 2016 Oct;36(10):1379-89. doi: 10.1007/s00296-016-3473-8. Epub 2016 Apr 7. PMID 27055444
- [Background] Mendonca ME, Simis M, Grecco LC, Battistella LR, Baptista AF, Fregni F. Transcranial Direct Current Stimulation Combined with Aerobic Exercise to Optimize Analgesic Responses in Fibromyalgia: A Randomized Placebo-Controlled Clinical Trial. Front Hum Neurosci. 2016 Mar 10;10:68. doi: 10.3389/fnhum.2016.00068. eCollection 2016. PMID 27014012
- [Background] Coppieters I, Cagnie B, Nijs J, van Oosterwijck J, Danneels L, De Pauw R, Meeus M. Effects of Stress and Relaxation on Central Pain Modulation in Chronic Whiplash and Fibromyalgia Patients Compared to Healthy Controls. Pain Physician. 2016 Mar;19(3):119-30. PMID 27008285
- [Background] Yuan SL, Matsutani LA, Marques AP. Effectiveness of different styles of massage therapy in fibromyalgia: a systematic review and meta-analysis. Man Ther. 2015 Apr;20(2):257-64. doi: 10.1016/j.math.2014.09.003. Epub 2014 Oct 5. PMID 25457196
- [Background] Liptan G, Mist S, Wright C, Arzt A, Jones KD. A pilot study of myofascial release therapy compared to Swedish massage in fibromyalgia. J Bodyw Mov Ther. 2013 Jul;17(3):365-70. doi: 10.1016/j.jbmt.2012.11.010. Epub 2013 Jan 3. PMID 23768283
- [Background] Castro-Sanchez AM, Mataran-Penarrocha GA, Arroyo-Morales M, Saavedra-Hernandez M, Fernandez-Sola C, Moreno-Lorenzo C. Effects of myofascial release techniques on pain, physical function, and postural stability in patients with fibromyalgia: a randomized controlled trial. Clin Rehabil. 2011 Sep;25(9):800-13. doi: 10.1177/0269215511399476. Epub 2011 Jun 14. PMID 21673013
- [Background] Castro-Sanchez AM, Mataran-Penarrocha GA, Granero-Molina J, Aguilera-Manrique G, Quesada-Rubio JM, Moreno-Lorenzo C. Benefits of massage-myofascial release therapy on pain, anxiety, quality of sleep, depression, and quality of life in patients with fibromyalgia. Evid Based Complement Alternat Med. 2011;2011:561753. doi: 10.1155/2011/561753. Epub 2010 Dec 28. PMID 21234327
- [Background] Ericsson A, Palstam A, Larsson A, Lofgren M, Bileviciute-Ljungar I, Bjersing J, Gerdle B, Kosek E, Mannerkorpi K. Resistance exercise improves physical fatigue in women with fibromyalgia: a randomized controlled trial. Arthritis Res Ther. 2016 Jul 30;18:176. doi: 10.1186/s13075-016-1073-3. PMID 27473164